CLINICAL TRIAL: NCT07302763
Title: Four-Timepoint Multi-tracer PET Imaging to Characterize Metastatic prOstate Cancer Heterogeneity
Acronym: 4TMPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frederic Pouliot (Other)
Responsible Party: Sponsor-Investigator, Frederic Pouliot, Principal Investigator, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-7376
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: mCRPC (Metastatic Castration-resistant Prostate Cancer)
Keywords: oncology; molecular imaging tracers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET with FDG, PSMA and DOTATATE (Experimental)
  Interventions: Diagnostic Test: PET Tracer

INTERVENTIONS:
Diagnostic Test: PET Tracer — Multi-tracer PET imaging to characterize metastatic prOstate Cancer heterogeneity

SUMMARY:
Imaging modalities currently used in the clinics do not image cancer, but the effect ofncancer on bone (bone scan) or on the anatomy (CT-scan). Bone scan and CT-scan are therefore named conventional imaging (CI) modalities. Positron Emission Tomography (PET) is an imaging technique that uses tracers to measure cancer activity in each lesion and is therefore quantitative. Usually, treatment changes in metastatic prostate cancers are based on the appearance of new lesions on CI, named metastases. Prostate cancer metastases have been shown to be clonal, which means that there are several cancers within each patient, potentially with divergent behaviors under therapy. In other words, some metastases might be resistant to a systemic therapy like chemotherapy, while others might be sensitive. The study proposes here to use molecular imaging by positron emission tomography to image and quantify the activity of prostate cancer cells in each metastasis before start, after 3 months and after progression during systemic therapy.

Each metastasis will then be measured to assess whether there is an increase (resistance) or a decrease (response) in prostate cancer cell activity. The analysis will determine how many metastases progress or remain stable when new metastases appear on conventional imaging (polyclonal resistance), as well as the impact of a change in therapy on metastases that were previously stable when cancer progressed elsewhere. In addition, the genes expressed in responding and non-responding metastases will be analyzed to identify gene expression patterns associated with resistance and/or response. Overall, this study aims to characterize metastatic prostate cancer clonal resistance mechanisms using serial PET molecular imaging and imaging-guided genomics.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single-arm, non-randomized study using a multi-timepoint triple tracer molecular imaging to characterize intra-patient cancer phenotypes between metastases and to monitor phenotypic plasticity non-invasively. This will be done using 18F-FDG, 68Ga-PSMA (or any other PSMA tracer) and 68Ga-DOTATATE in participants progressing with CRPC and showing at least 3 metastases after conventional imaging. Any PSMA tracer could be used but the first PSMA-PET scan determines the PSMA radiotracer that will be used throughout the study, in order to make the analysis of the radiographic evolution of metastases more accurate (e.g. 68Ga-PSMA-617 or 18F-DCF-PyL or 68Ga-PSMA-11). The reference imaging must have been performed either: 1) after biochemical progression on treatment OR 2) at least 90 days after last treatment has begun if imaging was performed while patient was still responding (to avoid disappearance of metastasis due to treatment response). These imaging will include: 1) bone scan or 18F-Na-PET/CT AND either chest/abdomen CT or chest CT and abdomen MRI OR 2) 18F-FDG-PET/CT. This study is planned to be conducted in up to 4 sites in Canada. Eligible participants (see Section for Eligibility Criteria) will be enrolled in a non-randomized, sequential manner, with competitive enrollment between study sites. A total of 45 participants will be accrued. Enrolled participants will undergo 18F-FDG, 68Ga- or 18F-PSMA and 68Ga-DOTATATE-PET/CT scans. After initial triple tracer PET molecular imaging, the participants will be treated with cabazitaxel or docetaxel or ARPI (as standard of care or as an investigational agent) or PSMA-radioligand therapy (as standard of care or as an investigational agent). Three (3) months after initiation of systemic therapy double-tracer (PSMA & FDG) PET/CT imaging will be performed. Participants will continue their therapy and once progression will occur (V3, Progression 1), triple tracer will be repeated and a biopsy of a progressive lesion will be executed. Patients will be treated with a mandatory second line of approved mCRPC systemic therapies: PSMA-RLT therapy (Pluvicto 177Lu-PSMA-617) or Olaparib (PARPi) if they are found with homologous recombination repair (HRR) mutation (a predictive biomarker for PARPi). If not HRR mutated nor eligible to PSMA-RLT, a second line of approved mCRPC systemic therapy or research protocol will be offered. At Progression 2 (V4) (after treatment change following Progression 1), double-tracer 68Ga-PSMA and 18F-FDG PET/CT imaging will be repeated (DOTATATE scan will be optional). The patient will have another biopsy of a progressing lesion and an optional second biopsy of a non-progressing site offered.

ELIGIBILITY:
Inclusion Criteria:

1. Assign male at birth, any gender ≥ 18 years old;
2. Histologically or cytologically proven adenocarcinoma of the prostate;
3. Metastatic disease documented by at least 3 metastatic active lesions*, ** on whole body bone scan and/or measurable soft tissue on CT-scan (lymph nodes and visceral lesions);
4. CRPC & post-androgen receptor pathway inhibitor (ARPI) defined by progression under continuous castration (measured serum testosterone ≤50 ng/dL [1.73 nM]) AND an ARPI (darolutamide, apalutamide, enzalutamide or abiraterone acetate);
5. Eligible for taxane chemotherapy or PSMA-radioligand therapy (before imaging); 6-Able and willing to provide signed informed consent and to comply with protocol requirements.

   * Metastatic lesions on imaging are defined either: ≥ 10 mm on CT scan or caliper (for lymph nodes, see below), ≥ 20 mm on chest X-ray, lymph node ≥ 10 mm or having grown by ≥ 5 mm from baseline CT, any metastasis described on bone scan counts as a lesion. Of note: A bone lesion that has been treated by radiation is excluded from the lesions counted in the criterion of ≥ 3 lesions.

     * The reference imaging (scan with 3 metastases) confirming eligibility must be done either: 1) after biochemical progression on treatment OR 2) ≥ 90 days after last treatment has begun if imaging was performed while patient was still responding (to avoid disappearance of metastasis due to response).

Exclusion Criteria:

* 1. Another non-cutaneous malignancy or melanoma diagnosed in the past 5 years; 2. Currently under a randomized controlled trial with unknown allocation; 3-Any disease or condition limiting the patient's capacity to execute the study procedures, based on the investigators' opinion;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the change in prevalence of IIH of mCRPC undergoing consecutive lines of systemic therapy. | At Baseline and at the date of first and second documented progression, assessed up to 60 months
  Percentage of patients that show heterogeneous FDG and PSMA tracer uptakes between at least two metastases at baseline and at each progression following consecutive lines1 of study systemic therapies.
Determine intrapatient intermetastasis therapeutic heterogeneous response (IIHR) in mCRPC patients. | At the date of first and second documented progression, assessed up to 60 months
  Percentage of patients that show opposite FDG and/or PSMA tracer uptake and/or ratio responses between two metastases after first and second study systemic therapy.

SECONDARY OUTCOMES:
Evaluate the impact of systemic treatment change on progressing and non-progressing FDG or PSMA PET lesions under last treatment. | At the date of first and second documented progression, assessed up to 60 months
  Percentage of metastases per patient that will show a significant increase or decrease of FDG or PSMA tracer uptake or ratio after subsequent treatment change for progression.
Correlate histopathology of biopsies to imaging phenotypes. | At the date of first and second documented progression, assessed up to 60 months
  Associate histopathology and immunohistochemistry (IHC) with double tracer imaging phenotypes of biopsied patients.

OTHER OUTCOMES:
Link radiomic, and genomic features of single-timepoint and sequential multitracer PET imaging with clinical outcomes. Characterize the biological features of FDG positive/DOTATATE any/PSMA negative lesions (poor prognosis) vs PSMA positive/FDG any/DO | At the date of randomization, then 3 months after randomizaton and at the date of first and second documented progression, assessed up to 60 months
  1. Molecular imaging parameters (including DOTATATE data) and genomics that will predict radiographic or clinical failure to systemic therapy from data at baseline, 3 months and at progression.
  2. Molecular characterization of aggressive and less aggressive cancer by fresh frozen analysis (omics) and organoid cultures harvested from corresponding lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Pouliot, MD, PhD, Principal Investigator — CHU de Québec-Université Laval
Locations (1):
- CHU de Québec-Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No